CLINICAL TRIAL: NCT02473757
Title: Gene Therapy Follow up Protocol for Subjects Previously Enrolled in CAR T-Cell Studies
Brief Title: Gene Therapy Follow-up Protocol for People Previously Enrolled in CAR-T Cell Studies
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150141; 15-C-0141
Record Dates: First submitted 2015-06-13; First posted 2015-06-17 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11-26

CONDITIONS: Lyphoma, B-Cell; Leukemia, B-cell; Multiple Myeloma; Hematologic Malignancies
Keywords: Recombinant DNA Product; Laboratory Evaluation; NIH Office of Biotechnology Activities; Gamma-Retroviral Vectors; Natural History
MeSH Terms: conditions — Leukemia, B-Cell; Multiple Myeloma; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Cohort 1: Subjects who have received treatment on an NCI Surgery Branch CAR T-cell gene therapy protocols.

SUMMARY:
Background:

- Gene therapy is a way to treat or prevent disease using genes. It is monitored very closely by regulators because there can be long-term, unexpected side effects. NIH is required to try to contact people who have been treated with gene therapy at least annually for up to 15 years. This is to see if they have had any bad side effects. This trial does not include any therapy and is only for patients previously treated on gene-therapy trials at the NCI Surgery Branch who are no longer enrolled on their original gene therapy clinical trial.

Objective:

- To collect of long-term follow-up data on people who have been in gene transfer studies. This follow-up is required by regulators.

Eligibility:

- People age 18 and older who have been in a previous NCI Surgery Branch gene therapy research study.

Design:

* After they get the genetically modified cells, participants will:
* Have blood drawn 3, 6, and 12 months later.
* Have an annual clinic visit for the next 4 years. They will have a physical exam. They will answer questions about any signs of neurological, autoimmune, or blood disorders, or any new cancers. Blood may be drawn.
* Be called or emailed annually for the next 10 years. They will answer health questions. Blood samples may need to be taken.
* Participants will be asked for their current address and phone number. They will also be asked for the address and phone number of 1 or 2 people who will know their whereabouts. One of these should be a family member if possible,
* At the time of the participant s death, researchers will request permission from their family for an autopsy.

DETAILED DESCRIPTION:
Background:

-The National Cancer Institute Surgery Branch (NCI-SB) Branch investigator conducts clinical trials utilizing gene transfer. The current U.S. Food and Drug Administration (FDA) requirements for long term follow up may be up to fifteen years for some products. As this time period is frequently longer than studies are expected to be open, a long-term follow-up protocol is necessary to ensure the follow up of these subjects

Objectives:

-To facilitate collection of long term, follow up information on subjects who have participated in gene transfer studies as required by the U.S. Food and Drug Administration and other regulatory groups

Eligibility:

-Enrollment on a CAR T-cell treatment protocol for gene therapy.

Design:

-Patients will undergo physical exams; laboratory evaluation or phone follow up as required by the treatment protocol and/or as clinically indicated.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects who have received treatment on a CAR T-cell gene therapy protocol. Age >= 18 years as children are generally excluded from CAR T-cell gene therapy studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To facilitate collection of long term follow up information on subjects who have participated in gene transfer studies as required by the U.S. Food and Drug Administration and other regulatory groups
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09-24 (Actual); Primary Completion 2034-07-01 (Estimated); Study Completion 2050-08-01 (Estimated)

PRIMARY OUTCOMES:
To provide long term follow up of patients previously enrolled on treatment protocols in the NCI ETIB Branch. | 15 years
  List of long time adverse event frequency after Gene therapy drug

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-C-0141.html